CLINICAL TRIAL: NCT01443988
Title: A Prospective, Randomized Evaluation of Subjects With Open-angle Glaucoma, Pseudoexfoliative Glaucoma, or Ocular Hypertension Naïve to Medical and Surgical Therapy, Treated With Two Trabecular Micro-bypass Stents (iStent) or Travoprost Ophthalmic Solution 0.004%
Brief Title: Subjects With Open-angle Glaucoma, Pseudoexfoliative Glaucoma, or Ocular Hypertension Naïve to Medical and Surgical Therapy, Treated With Two Trabecular Micro-bypass Stents (iStent)or Travoprost
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCF-022
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Open-angle Glaucoma
Keywords: Open angle glaucoma; POAG; Ocular hypertension; Pseudoexfoliative glaucoma; Naïve to treatment
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iStent (Active Comparator): Implantation of two iStent devices
  Interventions: Device: iStent
- Drug (Active Comparator): Travoprost drops
  Interventions: Drug: Travoprost

INTERVENTIONS:
Device: iStent — Implantation of two iStent devices
  Arms: iStent
Drug: Travoprost — Travoprost drops
  Arms: Drug

SUMMARY:
Evaluation of the intraocular pressure (IOP) lowering effect of two iStent devices versus medical therapy in eyes of subjects with primary open-angle glaucoma, pseudoexfoliative glaucoma, or ocular hypertension naïve to medical and surgical therapy.

DETAILED DESCRIPTION:
Evaluation of the intraocular pressure (IOP) lowering effect of two iStent devices versus medical therapy in eyes of subjects with primary open-angle glaucoma, pseudoexfoliative glaucoma, or ocular hypertension naïve to medical and surgical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Phakic study eye
* IOP ≥ 21 mmHg and ≤ 40 mmHg at screening exam (OHT requires second screening)

Exclusion Criteria:

* Aphakic or pseudophakic eyes (AC-IOLs or PC-IOLs)
* Previous usage of topical prostaglandin analogues or prior medical therapy for glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change from screening in mean diurnal IOP (mm Hg) at the Month 12 visit. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lilit A Voskanyan, MD, PhD, Principal Investigator — S.V. Malayan Ophthalmological Center, Yerevan, Armenia
Locations (1):
- S.V. Malayan Ophthalmological Center, Yerevan, Armenia

REFERENCES:
- [Background] Vold SD, Voskanyan L, Tetz M, Auffarth G, Masood I, Au L, Ahmed II, Saheb H. Newly Diagnosed Primary Open-Angle Glaucoma Randomized to 2 Trabecular Bypass Stents or Prostaglandin: Outcomes Through 36 Months. Ophthalmol Ther. 2016 Dec;5(2):161-172. doi: 10.1007/s40123-016-0065-3. Epub 2016 Sep 12. PMID 27619225